CLINICAL TRIAL: NCT04127877
Title: Regional Electric Bio Impedance-assisted Monitoring of Cardiac, Vascular Resistance and Fluid Balance, in Chronic Hemodialysis Patients
Brief Title: Bio Impedance-assisted Monitoring of Chronic Hemodialysis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Principal Investigator, Adi Leiba, Proffesor Adi Leiba, head, Nephrology and Hypertension Institute,, Assuta Ashdod Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0069-18
Record Dates: First submitted 2019-10-13; First posted 2019-10-16 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Chronic Kidney Diseases; Hemodialysis Complication
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHRONIC HEMODIALYSIS PATIENTS, NICAS-ASSISTED MONITORING (Experimental): Chronic hemodialysis patients, NICAS-assisted monitored
  Interventions: Device: NICAS
- Control hemodialysis patients (No Intervention): Chronic hemodialysis patients, conventional clinical care and monitoring.

INTERVENTIONS:
Device: NICAS — Electric regional bio impedance device
  Arms: CHRONIC HEMODIALYSIS PATIENTS, NICAS-ASSISTED MONITORING

SUMMARY:
Hemodynamic trends will be assessed using the device, in 100 dialysis sessions in 30 patients, who are prone to develop hypotensive episode during dialysis. Sitting blood pressures will be measured immediately prior to each hemodynamic measurement: before initiation of dialysis, every each hour and in the beginning of hypotension episode, just before the end and 10 min after the end of the treatment.

Gender, age, height, weight, electrode location and blood pressure data will be entered into the device. The device will measure and calculate hemodynamic parameters on each heart beat during 60 s and provides the averaged parameters.

Technology for hemodynamic measurements:

The device (NICaS, NI Medical) is a noninvasive regional bioimpedance cardiac measurement and analysis system (FDA 510k clearance no. K080941, 12 June 2009). The US Food and Drug Administration indication for use of the device states 'NICaS is intended to monitor and display hemodynamic parameters in males and females with known or suspected cardiac disorders needing cardiac assessment'.

SV will be measured by applying an alternating electrical current of 1.4mA at 30 kHz frequency through the patient's body via two pairs of tetrapolar sensors, one pair placed on the wrist of the nonaccess arm above the radial pulse and the other pair on the contralateral ankle above the posterior tibial pulse (Figure 1).

Figure 1 : Sensor location

SV is calculated by Frinerman's formula:

SV¼(dR/R) - q - (L2/Ri) - (ab)/b - KW - HF [2-4], where dR is the impedance change in the arterial system as a result of intraarterial expansion during systole, R is basal resistance, q is blood electrical resistance, L is the patient's height, Ri is basal resistance corrected for gender and age, KWis the correction of weight according to ideal values, HF is a hydration factor that takes into account the ratio between R and body mass index (BMI), which is correlated to body water volume, ab is the electrocardiogram (ECG) R-R wave interval and b is the diastolic time interval. SV is automatically calculated every 20 s and is the average of three measurements obtained consecutively during 60 s of monitoring. The SV index is calculated as SV/body surface area using the Du Bois formula [11]. Heart rate is calculated from a one channel ECG and cardiac (output) index¼SV index - heart rate/1000. Using an oscillometric method, sitting systolic and diastolic blood pressure measurements were made automatically by the dialysis machine. Mean arterial pressure [2 - (diastolicsystolic)/3], cardiac power index [CPI; mean arterial pressure (MAP) -cardiac index - 0.0022 w/m2; normal range 0.45-0.85w/m2] [12, 13] and total peripheral resistance (MAP/ cardiac index - 80 dyn - s/cm5 - m2; normal range 1600-3000 dyn - s/cm5- m2) [13] will be calculated.

As the device measures pulsatile flow and is blinded to constant flow, fluid removal during dialysis has no impact on measurement accuracy. This was recently validated by correlating SV to ECG measurements during hemodialysis treatments. Good correlation was maintained during treatment. Further, NICaS performance immunity to fluid reduction was demonstrated by the maintenance of correlation to ECG results throughout dialysis treatments [9]. The results are drawn on hemodynamic graphs showing the MAP (y-axis) as a function of cardiac index (x-axis); curves of total peripheral resistance index (TPRI) and CPI are displayed. Ranges for the normal population are depicted by a dotted octagon.

DETAILED DESCRIPTION:
Hemodynamic trends will be assessed using the device, in 100 dialysis sessions in 30 patients, who are prone to develop hypotensive episode during dialysis. Sitting blood pressures will be measured immediately prior to each hemodynamic measurement: before initiation of dialysis, every each hour and in the beginning of hypotension episode, just before the end and 10 min after the end of the treatment.

Gender, age, height, weight, electrode location and blood pressure data will be entered into the device. The device will measure and calculate hemodynamic parameters on each heart beat during 60 s and provides the averaged parameters.

Technology for hemodynamic measurements:

The device (NICaS, NI Medical) is a noninvasive regional bioimpedance cardiac measurement and analysis system (FDA 510k clearance no. K080941, 12 June 2009). The US Food and Drug Administration indication for use of the device states 'NICaS is intended to monitor and display hemodynamic parameters in males and females with known or suspected cardiac disorders needing cardiac assessment'.

SV will be measured by applying an alternating electrical current of 1.4mA at 30 kHz frequency through the patient's body via two pairs of tetrapolar sensors, one pair placed on the wrist of the nonaccess arm above the radial pulse and the other pair on the contralateral ankle above the posterior tibial pulse (Figure 1).

Figure 1 : Sensor location

SV is calculated by Frinerman's formula:

SV¼(dR/R) - q - (L2/Ri) - (ab)/b - KW - HF [2-4], where dR is the impedance change in the arterial system as a result of intraarterial expansion during systole, R is basal resistance, q is blood electrical resistance, L is the patient's height, Ri is basal resistance corrected for gender and age, KWis the correction of weight according to ideal values, HF is a hydration factor that takes into account the ratio between R and body mass index (BMI), which is correlated to body water volume, ab is the electrocardiogram (ECG) R-R wave interval and b is the diastolic time interval. SV is automatically calculated every 20 s and is the average of three measurements obtained consecutively during 60 s of monitoring. The SV index is calculated as SV/body surface area using the Du Bois formula [11]. Heart rate is calculated from a one channel ECG and cardiac (output) index¼SV index - heart rate/1000. Using an oscillometric method, sitting systolic and diastolic blood pressure measurements were made automatically by the dialysis machine. Mean arterial pressure [2 - (diastolicsystolic)/3], cardiac power index [CPI; mean arterial pressure (MAP) -cardiac index - 0.0022 w/m2; normal range 0.45-0.85w/m2] [12, 13] and total peripheral resistance (MAP/ cardiac index - 80 dyn - s/cm5 - m2; normal range 1600-3000 dyn - s/cm5- m2) [13] will be calculated.

As the device measures pulsatile flow and is blinded to constant flow, fluid removal during dialysis has no impact on measurement accuracy. This was recently validated by correlating SV to ECG measurements during hemodialysis treatments. Good correlation was maintained during treatment. Further, NICaS performance immunity to fluid reduction was demonstrated by the maintenance of correlation to ECG results throughout dialysis treatments [9]. The results are drawn on hemodynamic graphs showing the MAP (y-axis) as a function of cardiac index (x-axis); curves of total peripheral resistance index (TPRI) and CPI are displayed. Ranges for the normal population are depicted by a dotted octagon.

ELIGIBILITY:
Inclusion Criteria:

-Chronic hemodialysis patients

Exclusion Criteria:

* Age limits

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-18 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic adverse events | One year
  Extreme blood pressure decrease, hospitalization, death

CONTACTS AND LOCATIONS:
Overall Officials: Adi Leiba, Prof, Principal Investigator — ASSUTA HOSPITAL ASHDOD
Locations (1):
- Nephrology and Hypertention Institute, hemodialysis unit, Ashdod, Israel

IPD SHARING:
Plan to Share IPD: No